CLINICAL TRIAL: NCT01051349
Title: A Multicenter, Open-label, Extension Study to Evaluate the Long Term Safety and Efficacy of Daclizumab High Yield Process (DAC HYP) Monotherapy in Subjects With Multiple Sclerosis Who Have Completed Treatment in Study 205MS202 (SELECTION)
Brief Title: Safety and Efficacy Extension Study of Daclizumab High Yield Process (DAC HYP) (BIIB019) in Participants Who Have Completed Study 205MS202 (NCT00870740) to Treat Relapsing Remitting Multiple Sclerosis
Acronym: SELECTED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205-MS-203; 2009-015318-23 (EudraCT Number)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Daclizumab; daclizumab HYP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIIB019 (Experimental): Participants received BIIB019, 150 mg subcutaneous injection every 4 weeks up to Week 288.
  Interventions: Biological: BIIB019 (Daclizumab); Biological: trivalent seasonal influenza vaccine

INTERVENTIONS:
Biological: BIIB019 (Daclizumab) — Administered as specified in the treatment arm.
  Other Names: Daclizumab High Yield Process; DAC HYP
Biological: trivalent seasonal influenza vaccine — All participants who participate in the 2013-2014 influenza vaccine substudy will receive the vaccine at the study site

SUMMARY:
Primary Objective is to assess the safety of extended treatment with Daclizumab High Yield Process (DAC HYP, BIIB019) monotherapy in participants with relapsing remitting multiple sclerosis (RRMS). Secondary Objective is to assess the long-term immunogenicity of DAC HYP and to assess the durability of response to DAC HYP in preventing multiple sclerosis (MS) relapse, slowing disability progression, and reducing new MS lesion formation in this study population.

DETAILED DESCRIPTION:
This study will provide participants who complete Study 205MS202 (NCT00870740) with the option to receive continued open-label Daclizumab High Yield Process (DAC HYP) monotherapy and to evaluate the long-term safety, efficacy, and immunogenicity of DAC HYP monotherapy in participants with relapsing remitting multiple sclerosis (RRMS). Approximately 60 to 100 participants will be enrolled into an optional open-label, 16-week autoinjector substudy at a selected subset of sites which will run concurrently during the main study, and will evaluate the systemic exposure and local tolerability of subcutaneous administration of DAC HYP by autoinjector. The 2013-2014 trivalent influenza vaccine will be offered to all eligible participants as an optional substudy to assess the effect of DAC-HYP treatment on the immune response to vaccination,

ELIGIBILITY:
Main Study Eligibility:

Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Subjects who have completed 52 weeks in Study 205MS202 (NCT00870740) and were compliant with the 205MS202 protocol in the opinion of the Investigator.
* Women of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 4 months after their last dose of study treatment.

Key Exclusion Criteria:

* Subjects with any significant change in their medical status from the previous study that would prelude administration of Daclizumab High Yield Process (DAC HYP) as determined by the Investigator including laboratory tests or a current clinically significant condition that, in the opinion of the Investigator, would have excluded the subject's participation in the 205MS201 (NCT00390221) or 205MS202 (NCT00870740) studies. The Investigator must re-review the subject's medical fitness for participation and must consider any diseases that would preclude treatment.
* Any subject who has permanently discontinued study treatment in Study 205MS202 (NCT00870740) due to an adverse event.
* Current enrollment in any investigational drug study other than Study 205MS202 (NCT00870740).
* Ongoing treatment with any approved or experimental disease-modifying treatment for multiple sclerosis.
* For subjects currently taking valproic acid, carbamazepine, lamotrigine, or phenytoin:

  * Subjects treated with any of these agents for fewer than 6 months prior to study entry are excluded from study participation unless they discontinue the agent(s) prior to study entry.
  * Subjects treated with 2 or more of these agents for more than 6 months prior to study entry are excluded from study participation unless they reduce to ≤1 agent prior to study entry.
  * Subjects who have had dose escalations of one of these agents within the 6 months prior to study entry are excluded from study participation unless they revert to a previous dose that had been used for at least 6 months prior to study entry or unless they discontinue the agent prior to study entry
* Subjects who are currently receiving treatment with isoniazid, propylthiouracil, or nimesulide at the time of study entry and are not able to discontinue the agent or change to an alternative medication allowed by the protocol.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 410 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2016-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (52):
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Teplice
- Germany (4):
  - Research Site, Bayreuth
  - Research Site, Erlangen
  - Research Site, Marburg
  - Research Site, Rostock
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Siófok
- India (5):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Rajasthan
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Russia (11):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Smolensk
  - Research Site, Ufa
  - Research Site, Yaroskavi
- Ukraine (8):
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Poltava
  - Research Site, Zaporizhia
- United Kingdom (5):
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Gold R, Radue EW, Giovannoni G, Selmaj K, Havrdova EK, Montalban X, Stefoski D, Sprenger T, Robinson RR, Fam S, Smith J, Chalkias S, Giannattasio G, Lima G, Castro-Borrero W. Long-term safety and efficacy of daclizumab beta in relapsing-remitting multiple sclerosis: 6-year results from the SELECTED open-label extension study. J Neurol. 2020 Oct;267(10):2851-2864. doi: 10.1007/s00415-020-09835-y. Epub 2020 May 25. PMID 32451615
- [Derived] Gold R, Radue EW, Giovannoni G, Selmaj K, Havrdova E, Stefoski D, Sprenger T, Montalban X, Cohan S, Umans K, Greenberg SJ, Ozen G, Elkins J. Safety and efficacy of daclizumab in relapsing-remitting multiple sclerosis: 3-year results from the SELECTED open-label extension study. BMC Neurol. 2016 Jul 26;16:117. doi: 10.1186/s12883-016-0635-y. PMID 27461166
- [Derived] Gold R, Stefoski D, Selmaj K, Havrdova E, Hurst C, Holman J, Tornesi B, Akella S, McCroskery P. Pregnancy Experience: Nonclinical Studies and Pregnancy Outcomes in the Daclizumab Clinical Study Program. Neurol Ther. 2016 Dec;5(2):169-182. doi: 10.1007/s40120-016-0048-2. Epub 2016 Jul 13. PMID 27411694
- See also: The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS their families and healthcare providers — http://www.nationalmssociety.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 410 enrolled participants, 60 participants who received at least 6 consecutive monthly doses of DAC HYP in this study and had provided written informed consent were enrolled in to the autoinjector substudy and 91 participants who received seasonal trivalent influenza vaccine were enrolled in vaccine substudy (exploratory analyses).
Groups:
- BIIB019: Participants received BIIB019, 150 mg subcutaneous injection every 4 weeks up to Week 276.
Period: Overall Study
Arm/Group | BIIB019
Started | 410
Completed | 237
Not Completed | 173
Not completed — Adverse Event | 88
Not completed — Consent Withdrawn | 54
Not completed — Investigator Decision | 6
Not completed — Lost to Follow-up | 6
Not completed — Subject non-compliance | 7
Not completed — Reason not Specified | 12

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least 1 dose of study drug.
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254
  Male | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuation Due to AEs, Withdrawals Due to AEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Baseline up to 24 weeks after last dose of treatment (Up to 300 weeks)
Population: Safety population included participants who provided informed consent and received at least 1 dose of DAC HYP during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Participants
  Number of participants with an AEs | 358
  Number of participants with SAEs | 148
  Participants discontinuing treatment due to AE | 91
  Participants withdrawing from study due to AE | 90

2. Primary Outcome: Area Under the Concentration-Time Curve Over the Dosing Interval (AUC0-t) After Dose 4 for Daclizumab
Time Frame: Day 90 (Week 12) at predose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14, 21 and 28 days post-dose
Population: Pharmacokinetic analysis population included all participants in the Autoinjector Substudy with a sufficient number of samples available for analysis by randomized treatment group.
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Groups:
- BIIB019 (Prefilled Syringe [PFS]): Participants received BIIB019, 150 mg subcutaneous injection in a prefilled syringe every 4 weeks up to Week 276.
- BIIB019 (Autoinjector [AI]): Participants received BIIB019, 150 mg subcutaneous injection using an autoinjector every 4 weeks up to Week 276.
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
hr*mg/mL | 610.5 (253.89) | 666.8 (253.19)

3. Secondary Outcome: Number of Participants With New or Newly Enlarging T2 Hyperintense Lesions Compared to Baseline
Description: New or newly enlarging T2 hyperintense lesions evaluated by magnetic resonance imaging (MRI) and analyzed by a central reader.
Time Frame: From Baseline through 288 weeks
Population: Intent-to-treat (ITT) population included participants who provided informed consent and received at least 1 dose of DAC HYP during the study. Here 'n' indicates number of participants who were evaluable at specific time points.
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Participants
  Week 48 New or newly enlarging T2 lesions=0: number analyzed (Participants) | 363
  Week 48 New or newly enlarging T2 lesions=0 | 255
  Week 48 New or newly enlarging T2 lesions=1: number analyzed (Participants) | 363
  Week 48 New or newly enlarging T2 lesions=1 | 39
  Week 48 New or newly enlarging T2 lesions=2: number analyzed (Participants) | 363
  Week 48 New or newly enlarging T2 lesions=2 | 27
  Week 48 New or newly enlarging T2 lesions=3: number analyzed (Participants) | 363
  Week 48 New or newly enlarging T2 lesions=3 | 12
  Week 48 New or newly enlarging T2 lesions=4: number analyzed (Participants) | 363
  Week 48 New or newly enlarging T2 lesions=4 | 5
  Week 48 New/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 363
  Week 48 New/newly enlarging T2 lesions=5-6 | 6
  Week 48 New/newly enlarging T2 lesions=7-10: number analyzed (Participants) | 363
  Week 48 New/newly enlarging T2 lesions=7-10 | 8
  Week 48 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 363
  Week 48 New/newly enlarging T2 lesions>=11 | 11
  Week 96 New/newly enlarging T2 lesions=0: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=0 | 213
  Week 96 New/newly enlarging T2 lesions=1: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=1 | 41
  Week 96 New/newly enlarging T2 lesions=2: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=2 | 17
  Week 96 New/newly enlarging T2 lesions=3: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=3 | 17
  Week 96 New/newly enlarging T2 lesions=4: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=4 | 11
  Week 96 New/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=5-6 | 6
  Week 96 New/newly enlarging T2 lesions=7-10: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions=7-10 | 10
  Week 96 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 333
  Week 96 New/newly enlarging T2 lesions>=11 | 18
  Week 144 New/newly enlarging T2 lesions=0: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=0 | 33
  Week 144 New/newly enlarging T2 lesions=1: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=1 | 5
  Week 144 New/newly enlarging T2 lesions=2: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=2 | 1
  Week 144 New/newly enlarging T2 lesions=3: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=3 | 2
  Week 144 New/newly enlarging T2 lesions=4: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=4 | 1
  Week 144 New/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=5-6 | 4
  Week 144 New/newly enlarging T2 lesions=7-10: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions=7-10 | 1
  Week 144 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 53
  Week 144 New/newly enlarging T2 lesions>=11 | 6
  Week 192 New/newly enlarging T2 lesions=0: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions=0 | 144
  Week 192 New/newly enlarging T2 lesions=1: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions=1 | 30
  Week 192 New/newly enlarging T2 lesions=2: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions=2 | 24
  Week 192 New/newly enlarging T2 lesions=3: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions=3 | 13
  Week 192 New/newly enlarging T2 lesions=4: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions=4 | 9
  Week 192 Ne/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 262
  Week 192 Ne/newly enlarging T2 lesions=5-6 | 11
  Week 192 New/newly enlarging T2lesions=7-10: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2lesions=7-10 | 11
  Week 192 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 262
  Week 192 New/newly enlarging T2 lesions>=11 | 20
  Week 240 New/newly enlarging T2 lesions=0: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=0 | 60
  Week 240 New/newly enlarging T2 lesions=1: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=1 | 10
  Week 240 New/newly enlarging T2 lesions=2: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=2 | 14
  Week 240 New/newly enlarging T2 lesions=3: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=3 | 9
  Week 240 New/newly enlarging T2 lesions=4: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=4 | 7
  Week 240 New/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions=5-6 | 7
  Week 240 New/newly enlarging T2lesions=7-10: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2lesions=7-10 | 3
  Week 240 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 121
  Week 240 New/newly enlarging T2 lesions>=11 | 11
  Week 288 New/newly enlarging T2 lesions=0: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=0 | 14
  Week 288 New/newly enlarging T2 lesions=1: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=1 | 1
  Week 288 New/newly enlarging T2 lesions=2: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=2 | 4
  Week 288 New/ newly enlarging T2 lesions=3: number analyzed (Participants) | 27
  Week 288 New/ newly enlarging T2 lesions=3 | 1
  Week 288 New/newly enlarging T2 lesions=4: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=4 | 0
  Week 288 New/newly enlarging T2 lesions=5-6: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=5-6 | 1
  Week 288 New/newly enlarging T2 lesions=7-10: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions=7-10 | 3
  Week 288 New/newly enlarging T2 lesions>=11: number analyzed (Participants) | 27
  Week 288 New/newly enlarging T2 lesions>=11 | 3

4. Secondary Outcome: Annual Change in Volume of New or Newly Enlarging T2 Hyperintense Lesions Compared to Baseline
Description: New or newly enlarging T2 hyperintense lesions evaluated by MRI and analyzed by a central reader.
Time Frame: From Baseline through 288 weeks
Population: ITT population included participants who provided informed consent and received at least 1 dose of DAC HYP during the study. Here 'n' indicates number of participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | BIIB019
Number analyzed (Participants) | 410
mm^3
  Change from Baseline at Week 48: number analyzed (Participants) | 362
  Change from Baseline at Week 48 | -340.8 (1237.64)
  Change from Baseline at Week 96: number analyzed (Participants) | 330
  Change from Baseline at Week 96 | -237.7 (1382.86)
  Change from Baseline at Week 144: number analyzed (Participants) | 51
  Change from Baseline at Week 144 | 38.2 (1825.06)
  Change from Baseline at Week 192: number analyzed (Participants) | 262
  Change from Baseline at Week 192 | -251.2 (2326.41)
  Change from Baseline at Week 240: number analyzed (Participants) | 122
  Change from Baseline at Week 240 | -269.7 (1188.82)
  Change from Baseline at Week 288: number analyzed (Participants) | 27
  Change from Baseline at Week 288 | 31.9 (1008.87)

5. Secondary Outcome: Number of Participants With Total Number of New Gadolinium-enhancing Lesions
Description: New Gadolinium-enhancing lesions was evaluated by MRI and analyzed by a central reader.
Time Frame: From Baseline through 288 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Participants
  Week 48 new Gd-enhancing lesions=1: number analyzed (Participants) | 372
  Week 48 new Gd-enhancing lesions=1 | 22
  Week 48 new Gd-enhancing lesions=2: number analyzed (Participants) | 372
  Week 48 new Gd-enhancing lesions=2 | 3
  Week 48 new Gd-enhancing lesions=3: number analyzed (Participants) | 372
  Week 48 new Gd-enhancing lesions=3 | 6
  Week 48 new Gd-enhancing lesions=>4: number analyzed (Participants) | 372
  Week 48 new Gd-enhancing lesions=>4 | 11
  Week 96 new Gd-enhancing lesions=1: number analyzed (Participants) | 338
  Week 96 new Gd-enhancing lesions=1 | 14
  Week 96 new Gd-enhancing lesions=2: number analyzed (Participants) | 338
  Week 96 new Gd-enhancing lesions=2 | 7
  Week 96 new Gd-enhancing lesions=3: number analyzed (Participants) | 338
  Week 96 new Gd-enhancing lesions=3 | 4
  Week 96 new Gd-enhancing lesions=>4: number analyzed (Participants) | 338
  Week 96 new Gd-enhancing lesions=>4 | 5
  Week 144 new Gd-enhancing lesions=1: number analyzed (Participants) | 55
  Week 144 new Gd-enhancing lesions=1 | 1
  Week 144 new Gd-enhancing lesions=2: number analyzed (Participants) | 55
  Week 144 new Gd-enhancing lesions=2 | 0
  Week 144 new Gd-enhancing lesions=3: number analyzed (Participants) | 55
  Week 144 new Gd-enhancing lesions=3 | 1
  Week 144 new Gd-enhancing lesions=>4: number analyzed (Participants) | 55
  Week 144 new Gd-enhancing lesions=>4 | 2
  Week 192 new Gd-enhancing lesions=1: number analyzed (Participants) | 266
  Week 192 new Gd-enhancing lesions=1 | 13
  Week 192 new Gd-enhancing lesions=2: number analyzed (Participants) | 266
  Week 192 new Gd-enhancing lesions=2 | 5
  Week 192 new Gd-enhancing lesions=3: number analyzed (Participants) | 266
  Week 192 new Gd-enhancing lesions=3 | 1
  Week 192 new Gd-enhancing lesions=>4: number analyzed (Participants) | 266
  Week 192 new Gd-enhancing lesions=>4 | 0
  Week 240 new Gd-enhancing lesions=1: number analyzed (Participants) | 124
  Week 240 new Gd-enhancing lesions=1 | 5
  Week 240 new Gd-enhancing lesions=2: number analyzed (Participants) | 124
  Week 240 new Gd-enhancing lesions=2 | 0
  Week 240 new Gd-enhancing lesions=3: number analyzed (Participants) | 124
  Week 240 new Gd-enhancing lesions=3 | 0
  Week 240 new Gd-enhancing lesions=>4: number analyzed (Participants) | 124
  Week 240 new Gd-enhancing lesions=>4 | 0
  Week 288 new Gd-enhancing lesions=1: number analyzed (Participants) | 27
  Week 288 new Gd-enhancing lesions=1 | 2
  Week 288 new Gd-enhancing lesions=2: number analyzed (Participants) | 27
  Week 288 new Gd-enhancing lesions=2 | 0
  Week 288 new Gd-enhancing lesions=3: number analyzed (Participants) | 27
  Week 288 new Gd-enhancing lesions=3 | 0
  Week 288 new Gd-enhancing lesions=>4: number analyzed (Participants) | 27
  Week 288 new Gd-enhancing lesions=>4 | 0

6. Secondary Outcome: Annual Change in Number of T1 Hypointense Lesions
Time Frame: From Baseline through 288 weeks
Population: T1 hypointense lesions changes reflect tissue destruction. Volume of T1 hypointense lesions is deemed a more valuable assessment. Hence number of T1 hypointense lesions were not assessed and reported.
Arm/Group | BIIB019
Number analyzed (Participants) | 0

7. Secondary Outcome: Annual Change in Volume of New Gadolinium-Enhancing Lesions
Time Frame: From Baseline through 288 weeks
Population: Gd enhancing lesion volume reflects acute inflammatory activity. The number of Gd lesions is a more valuable outcome measure. Hence the volume of Gd enhancing lesions was not assessed and reported.
Arm/Group | BIIB019
Number analyzed (Participants) | 0

8. Secondary Outcome: Annual Change in Volume of T1 Hypointense Lesions
Description: Volume of T1 hypointense lesions was evaluated by MRI and analyzed by a central reader.
Time Frame: From Baseline through 288 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | BIIB019
Number analyzed (Participants) | 410
mm^3
  Change from Baseline at Week 48: number analyzed (Participants) | 360
  Change from Baseline at Week 48 | -183.5 (370.66)
  Change from Baseline at Week 96: number analyzed (Participants) | 325
  Change from Baseline at Week 96 | -160.6 (443.78)
  Change from Baseline at Week 144: number analyzed (Participants) | 51
  Change from Baseline at Week 144 | -142.4 (432.57)
  Change from Baseline at Week 192: number analyzed (Participants) | 259
  Change from Baseline at Week 192 | -115.2 (826.84)
  Change from Baseline at Week 240: number analyzed (Participants) | 121
  Change from Baseline at Week 240 | -140.8 (514.38)
  Change from Baseline at Week 288: number analyzed (Participants) | 27
  Change from Baseline at Week 288 | -148.4 (500.07)

9. Secondary Outcome: Percent Change in Total Brain Volume
Description: To assess brain atrophy, total brain volume was be measured by MRI and analyzed by a central reader.
Time Frame: From Baseline through 288 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BIIB019
Number analyzed (Participants) | 410
percent change
  Change from Week 0 to Week 48: number analyzed (Participants) | 347
  Change from Week 0 to Week 48 | -0.4 (1.00)
  Change from Week 48 to Week 96: number analyzed (Participants) | 303
  Change from Week 48 to Week 96 | -0.4 (0.78)
  Change from Week 96 to Week 144: number analyzed (Participants) | 37
  Change from Week 96 to Week 144 | -0.2 (1.00)
  Change from Week 144 to Week 192: number analyzed (Participants) | 30
  Change from Week 144 to Week 192 | -0.5 (0.59)
  Change from Week 192 to Week 240: number analyzed (Participants) | 86
  Change from Week 192 to Week 240 | -0.2 (0.83)
  Change from Week 240 to Week 288: number analyzed (Participants) | 27
  Change from Week 240 to Week 288 | 0.1 (0.73)

10. Secondary Outcome: Number of Participants With Antibodies to DAC HYP
Time Frame: Up to Week 288
Population: Safety population included participants who provided informed consent and received at least 1 dose of DAC HYP during the study. Here number of participants analyzed is the participants who were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 407
Participants | 43

11. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: Relapses are defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting at least 24 hours, and accompanied by new objective neurological findings upon examination by the Examining Neurologist. The ARR was calculated by tabulating the total number of relapses experienced in the group divided by the number of days up to the end of study, and the ratio then multiplied by 365. Adjusted ARR was reported.
Time Frame: Week 288
Population: ITT population included participants who provided informed consent and received at least 1 dose of DAC HYP during the study.
Measure: Number (95% Confidence Interval); unit: relapses per person-year
Arm/Group | BIIB019
Number analyzed (Participants) | 410
relapses per person-year | 0.124 [0.099 to 0.156]

12. Secondary Outcome: Number of Participants With Sustained Disability Progression for 12 Weeks
Description: Sustained disability progression defined by at least a 1.0-point increase on the Expanded Disability Status Scale (EDSS) from a baseline EDSS ≥1.0 that is sustained for 12 weeks, or at least a 1.5-point increase on the EDSS from a baseline EDSS <1.0 that is sustained for 12 weeks. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10, with higher scores indicating more disability.
Time Frame: Week 48 up to Week 288
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Participants
  Weeks 0 - 48 | 22
  Weeks 49 - 96 | 17
  Weeks 97 - 144 | 13
  Weeks 145 -192 | 7
  Week 193 - 288 | 2

13. Secondary Outcome: Number of Participants With Sustained Disability Progression for 24 Weeks
Description: Sustained disability progression defined by at least a 1.0-point increase on the Expanded Disability Status Scale (EDSS) from a baseline EDSS ≥1.0 that is sustained for 24 weeks, or at least a 1.5-point increase on the EDSS from a baseline EDSS <1.0 that is sustained for 24 weeks. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10, with higher scores indicating more disability.
Time Frame: Week 48 up to Week 288
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019
Number analyzed (Participants) | 410
Participants
  Weeks 0 - 48 | 19
  Weeks 49 - 96 | 18
  Weeks 97 - 144 | 11
  Weeks 145 -192 | 7
  Week 193 - 288 | 3

14. Secondary Outcome: Observed Maximum Concentration (Cmax) After Dose 4 for Daclizumab
Time Frame: Day 90 (Week 12) at predose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14, 21 and 28 days post-dose
Population: Pharmacokinetic analysis population included all participants with a sufficient number of samples available for analysis.
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- BIIB019 (Prefilled Syringe [PFS]): Participants received BIIB019, 150 mg subcutaneous injection in a prefilled syringe every 4 weeks up to Week 288.
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
mg/mL | 31.8 (13.11) | 33.6 (14.79)

15. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) for Daclizumab After Dose 4
Time Frame: Day 90 (Week 12) at predose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14, 21 and 28 days post-dose
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
hour | 5.0 [1 to 14] | 6.0 [1 to 14]

16. Secondary Outcome: Observed Minimum Concentration (Cmin) for Daclizumab After Dose 4
Time Frame: Day 90 (Week 12) at predose and 8, 24, 72 and 120 hours post-dose and 7, 10, 14, 21 and 28 days post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
mg/mL | 13.8 (7.13) | 15.7 (7.31)

17. Secondary Outcome: Participant-Reported Pain Visual Analog Scale (VAS) Score
Description: The VAS is a 10 cm-long horizontal line labeled with 2 extremes of pain at either end ("0 [no pain]" on the left and "100 [very painful]" on the right). The participant rates their perceived pain of each injection by placing a vertical mark on the line to indicate the level of pain.
Time Frame: First injection (Day 1) and fourth injection (Day 90) 0 hour, 30 minutes, 60 minutes and 8 hours post-dose
Population: The participants who were enrolled in auto-injector sub study were evaluated in this outcome measure. Here 'n' indicates number of participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
score on a scale
  First injection, 0 hour post-dose | 12.7 (17.45) | 14.5 (19.47)
  First injection, 30 minutes post-dose | 0.1 (0.31) | 0.4 (1.01)
  First injection, 60 minutes post-dose | 0.1 (0.25) | 0.3 (0.60)
  First injection, 8 hours post-dose | 0.1 (0.25) | 0.2 (0.50)
  Fourth injection, 0 hour post-dose: number analyzed (Participants) | 30 | 28
  Fourth injection, 0 hour post-dose | 14.5 (21.7) | 15.6 (24.70)
  Fourth injection, 30 minutes post-dose: number analyzed (Participants) | 30 | 28
  Fourth injection, 30 minutes post-dose | 0.9 (3.51) | 1.3 (3.42)
  Fourth injection, 60 minutes post-dose: number analyzed (Participants) | 30 | 28
  Fourth injection, 60 minutes post-dose | 0.0 (0.18) | 0.1 (0.31)
  Fourth injection, 8 hours post-dose: number analyzed (Participants) | 30 | 28
  Fourth injection, 8 hours post-dose | 0.1 (0.40) | 0.1 (0.31)

18. Secondary Outcome: Summary of Injection Site Assessment Performed by Clinician
Description: Injection site assessment was performed by clinician and are defined as erythema (redness) rated on a 4 point scale ranging from 0-3, where 0=none, 1=mild, 2=moderate and 3=severe; pigmentation changes (skin discoloration other than redness) rated on a 3 point scale from 0-2, where 0=none, 1=hypopigmentation and 2=hyperpigmentation; induration (swelling) rated on a 4 point scale ranging from 0-3, where 0=none, 1=mild, 2=moderate and 3=severe; tenderness to pressure rated on a 4 point scale ranging from 0-3, where 0=none, 1=mild, 2=moderate and 3=severe; and local temperature changes of injection sites rated on a 3 point scale where 0=normal, 1=warm and 1=hot. Only those score categories for which there was at least 1 participant are reported.
  Here, Injection=Inj, post-dose=PD
Time Frame: First injection (Day 1) and fourth injection (Day 90) 30 minutes; 8, 24, 72, and 120 hours; and 7, 10, and 14 days post-dose
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | BIIB019 (Prefilled Syringe [PFS]) | BIIB019 (Autoinjector [AI])
Number analyzed (Participants) | 30 | 30
Participants
  Erythema: Ist Inj 30 min PD: None | 29 | 29
  Erythema:Ist Inj 30 min PD: Mild | 1 | 1
  Erythema: Ist Inj 8 h PD: None | 30 | 29
  Erythema:Ist Inj 8 h PD: MIld | 0 | 1
  Erythema: Ist Inj 24 h PD: None: number analyzed (Participants) | 28 | 27
  Erythema: Ist Inj 24 h PD: None | 28 | 27
  Erythema: Ist Inj 72 h PD: None: number analyzed (Participants) | 26 | 26
  Erythema: Ist Inj 72 h PD: None | 26 | 26
  Erythema: Ist Inj 120 h PD: None: number analyzed (Participants) | 26 | 26
  Erythema: Ist Inj 120 h PD: None | 26 | 26
  Erythema: Ist Inj 7 days PD: None: number analyzed (Participants) | 26 | 26
  Erythema: Ist Inj 7 days PD: None | 26 | 26
  Erythema: Ist Inj 10 days PD: None: number analyzed (Participants) | 26 | 26
  Erythema: Ist Inj 10 days PD: None | 26 | 26
  Erythema: Ist Inj 14 days PD: None: number analyzed (Participants) | 26 | 26
  Erythema: Ist Inj 14 days PD: None | 26 | 26
  Erythema: 4th Inj 30 min PD: None | 30 | 28
  Erythema: 4th Inj 30 min PD: Mild: number analyzed (Participants) | 30 | 28
  Erythema: 4th Inj 30 min PD: Mild | 0 | 1
  Erythema: 4th Inj 8 h PD: None: number analyzed (Participants) | 30 | 28
  Erythema: 4th Inj 8 h PD: None | 30 | 28
  Erythema: 4th Inj 24 h PD: None: number analyzed (Participants) | 30 | 27
  Erythema: 4th Inj 24 h PD: None | 30 | 27
  Erythema: 4th Inj 72 h PD: None: number analyzed (Participants) | 29 | 26
  Erythema: 4th Inj 72 h PD: None | 29 | 26
  Erythema: 4th Inj 120 h PD: None: number analyzed (Participants) | 30 | 27
  Erythema: 4th Inj 120 h PD: None | 30 | 27
  Erythema: 4th Inj 7 days PD: None: number analyzed (Participants) | 30 | 28
  Erythema: 4th Inj 7 days PD: None | 30 | 28
  Erythema: 4th Inj 10 days PD: None: number analyzed (Participants) | 30 | 28
  Erythema: 4th Inj 10 days PD: None | 30 | 28
  Erythema: 4th Inj 14 days PD: None: number analyzed (Participants) | 30 | 28
  Erythema: 4th Inj 14 days PD: None | 30 | 28
  Pigmentation: 1st Inj, 30 min PD: None | 30 | 30
  Pigmentation: 1st Inj, 8 h PD: None | 30 | 30
  Pigmentation: 1st Inj, 24 h PD: None: number analyzed (Participants) | 28 | 27
  Pigmentation: 1st Inj, 24 h PD: None | 28 | 27
  Pigmentation: 1st Inj, 72 h PD: None: number analyzed (Participants) | 26 | 26
  Pigmentation: 1st Inj, 72 h PD: None | 26 | 26
  Pigmentation: 1st Inj, 120 h PD: None: number analyzed (Participants) | 26 | 26
  Pigmentation: 1st Inj, 120 h PD: None | 26 | 26
  Pigmentation: 1st Inj, 7 days PD: None: number analyzed (Participants) | 26 | 26
  Pigmentation: 1st Inj, 7 days PD: None | 26 | 26
  Pigmentation: 1st Inj, 10 days PD: None: number analyzed (Participants) | 26 | 26
  Pigmentation: 1st Inj, 10 days PD: None | 26 | 26
  Pigmentation: 1st Inj, 14 days PD: None: number analyzed (Participants) | 26 | 26
  Pigmentation: 1st Inj, 14 days PD: None | 26 | 26
  Pigmentation: 4th Inj, 30 min PD: None: number analyzed (Participants) | 30 | 28
  Pigmentation: 4th Inj, 30 min PD: None | 30 | 28
  Pigmentation: 4th Inj, 8 h PD: None: number analyzed (Participants) | 30 | 28
  Pigmentation: 4th Inj, 8 h PD: None | 30 | 28
  Pigmentation: 4th Inj, 24 h PD: None: number analyzed (Participants) | 30 | 27
  Pigmentation: 4th Inj, 24 h PD: None | 30 | 27
  Pigmentation: 4th Inj, 72 h PD: None: number analyzed (Participants) | 29 | 26
  Pigmentation: 4th Inj, 72 h PD: None | 28 | 26
  Pigmentation: 4th Inj, 72 h PD: Hyper-: number analyzed (Participants) | 29 | 26
  Pigmentation: 4th Inj, 72 h PD: Hyper- | 1 | 0
  Pigmentation: 4th Inj, 120 h PD: None: number analyzed (Participants) | 30 | 27
  Pigmentation: 4th Inj, 120 h PD: None | 29 | 27
  Pigmentation: 4th Inj, 120 h PD: Hyper-: number analyzed (Participants) | 30 | 27
  Pigmentation: 4th Inj, 120 h PD: Hyper- | 1 | 0
  Pigmentation: 4th Inj, 7 days PD: None: number analyzed (Participants) | 30 | 28
  Pigmentation: 4th Inj, 7 days PD: None | 30 | 28
  Pigmentation: 4th Inj, 10 days PD: None: number analyzed (Participants) | 30 | 28
  Pigmentation: 4th Inj, 10 days PD: None | 30 | 28
  Pigmentation: 4th Inj, 14 days PD: None: number analyzed (Participants) | 30 | 28
  Pigmentation: 4th Inj, 14 days PD: None | 30 | 28
  Induration: 1st Inj, 30 min PD: None | 30 | 30
  Induration: 1st Inj, 8 h PD: None | 30 | 30
  Induration: 1st Inj, 24 h PD: None: number analyzed (Participants) | 28 | 27
  Induration: 1st Inj, 24 h PD: None | 28 | 27
  Induration: 1st Inj, 72 h PD: None: number analyzed (Participants) | 26 | 26
  Induration: 1st Inj, 72 h PD: None | 26 | 26
  Induration: 1st Inj, 120 h PD: None: number analyzed (Participants) | 26 | 26
  Induration: 1st Inj, 120 h PD: None | 26 | 26
  Induration: 1st Inj, 7 days PD: None: number analyzed (Participants) | 26 | 26
  Induration: 1st Inj, 7 days PD: None | 26 | 26
  Induration: 1st Inj, 10 days PD: None: number analyzed (Participants) | 26 | 26
  Induration: 1st Inj, 10 days PD: None | 26 | 26
  Induration: 1st Inj, 14 days PD: None: number analyzed (Participants) | 26 | 26
  Induration: 1st Inj, 14 days PD: None | 26 | 26
  Induration: 4th Inj, 30 min PD: None (n=30, 28): number analyzed (Participants) | 30 | 28
  Induration: 4th Inj, 30 min PD: None (n=30, 28) | 30 | 28
  Induration: 4th Inj, 8 h PD: None: number analyzed (Participants) | 30 | 28
  Induration: 4th Inj, 8 h PD: None | 30 | 28
  Induration: 4th Inj, 24 h PD: None: number analyzed (Participants) | 30 | 27
  Induration: 4th Inj, 24 h PD: None | 30 | 27
  Induration: 4th Inj, 72 h PD: None: number analyzed (Participants) | 29 | 26
  Induration: 4th Inj, 72 h PD: None | 29 | 26
  Induration: 4th Inj, 120 h PD: None: number analyzed (Participants) | 30 | 27
  Induration: 4th Inj, 120 h PD: None | 30 | 27
  Induration: 4th Inj, 7 days PD: None: number analyzed (Participants) | 30 | 28
  Induration: 4th Inj, 7 days PD: None | 30 | 28
  Induration: 4th Inj, 10 days PD: None: number analyzed (Participants) | 30 | 28
  Induration: 4th Inj, 10 days PD: None | 30 | 28
  Induration: 4th Inj, 14 days PD: None: number analyzed (Participants) | 30 | 28
  Induration: 4th Inj, 14 days PD: None | 30 | 28
  Tenderness: 1st Inj, 30 min PD: None | 30 | 29
  Tenderness: 1st Inj, 30 min PD: Mild | 0 | 1
  Tenderness: 1st Inj, 8 h PD: None | 30 | 30
  Tenderness: 1st Inj, 24 h PD: None: number analyzed (Participants) | 28 | 27
  Tenderness: 1st Inj, 24 h PD: None | 28 | 27
  Tenderness: 1st Inj, 72 h PD: None: number analyzed (Participants) | 26 | 26
  Tenderness: 1st Inj, 72 h PD: None | 26 | 26
  Tenderness: 1st Inj, 120 h PD: None: number analyzed (Participants) | 26 | 26
  Tenderness: 1st Inj, 120 h PD: None | 26 | 26
  Tenderness: 1st Inj, 7 days PD: None: number analyzed (Participants) | 26 | 26
  Tenderness: 1st Inj, 7 days PD: None | 26 | 26
  Tenderness: 1st Inj, 10 days PD: None: number analyzed (Participants) | 26 | 26
  Tenderness: 1st Inj, 10 days PD: None | 26 | 26
  Tenderness: 1st Inj, 14 days PD: None: number analyzed (Participants) | 26 | 26
  Tenderness: 1st Inj, 14 days PD: None | 26 | 26
  Tenderness: 4th Inj, 30 min PD: None: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 30 min PD: None | 30 | 27
  Tenderness: 4th Inj, 30 min PD: Mild: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 30 min PD: Mild | 0 | 1
  Tenderness: 4th Inj, 8 h PD: None: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 8 h PD: None | 30 | 27
  Tenderness: 4th Inj, 8 h PD: Mild: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 8 h PD: Mild | 0 | 1
  Tenderness: 4th Inj, 24 h PD: None: number analyzed (Participants) | 30 | 27
  Tenderness: 4th Inj, 24 h PD: None | 30 | 27
  Tenderness: 4th Inj, 72 h PD: None: number analyzed (Participants) | 29 | 26
  Tenderness: 4th Inj, 72 h PD: None | 29 | 26
  Tenderness: 4th Inj, 120 h PD: None: number analyzed (Participants) | 30 | 27
  Tenderness: 4th Inj, 120 h PD: None | 30 | 27
  Tenderness: 4th Inj, 7 days PD: None: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 7 days PD: None | 30 | 28
  Tenderness: 4th Inj, 10 days PD: None: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 10 days PD: None | 30 | 28
  Tenderness: 4th Inj, 14 days PD: None: number analyzed (Participants) | 30 | 28
  Tenderness: 4th Inj, 14 days PD: None | 30 | 28
  Temperature: 1st Inj, 30 min PD: Normal | 30 | 30
  Temperature: 1st Inj, 8 h PD: Normal | 30 | 30
  Temperature: 1st Inj, 24 h PD: Normal: number analyzed (Participants) | 28 | 27
  Temperature: 1st Inj, 24 h PD: Normal | 28 | 27
  Temperature: 1st Inj, 72 h PD: Normal: number analyzed (Participants) | 26 | 26
  Temperature: 1st Inj, 72 h PD: Normal | 26 | 26
  Temperature: 1st Inj, 120 h PD: Normal: number analyzed (Participants) | 26 | 26
  Temperature: 1st Inj, 120 h PD: Normal | 26 | 26
  Temperature: 1st Inj, 7 days PD: Normal: number analyzed (Participants) | 26 | 26
  Temperature: 1st Inj, 7 days PD: Normal | 26 | 26
  Temperature: 1st Inj,10 days PD: Normal: number analyzed (Participants) | 26 | 26
  Temperature: 1st Inj,10 days PD: Normal | 26 | 26
  Temperature: 1st Inj,14 days PD: Normal: number analyzed (Participants) | 26 | 26
  Temperature: 1st Inj,14 days PD: Normal | 26 | 26
  Temperature: 4th Inj, 30 min PD: Normal: number analyzed (Participants) | 30 | 28
  Temperature: 4th Inj, 30 min PD: Normal | 30 | 28
  Temperature: 4th Inj, 8 h PD: Normal: number analyzed (Participants) | 30 | 28
  Temperature: 4th Inj, 8 h PD: Normal | 30 | 28
  Temperature: 4th Inj, 24 h PD: Normal: number analyzed (Participants) | 30 | 27
  Temperature: 4th Inj, 24 h PD: Normal | 30 | 27
  Temperature: 4th Inj, 72 h PD: Normal: number analyzed (Participants) | 29 | 26
  Temperature: 4th Inj, 72 h PD: Normal | 29 | 26
  Temperature: 4th Inj, 120 h PD: Normal: number analyzed (Participants) | 30 | 27
  Temperature: 4th Inj, 120 h PD: Normal | 30 | 27
  Temperature: 4th Inj, 7 days PD: Normal: number analyzed (Participants) | 30 | 28
  Temperature: 4th Inj, 7 days PD: Normal | 30 | 28
  Temperature: 4th Inj,10 days PD: Normal: number analyzed (Participants) | 30 | 28
  Temperature: 4th Inj,10 days PD: Normal | 30 | 28
  Temperature: 4th Inj,14 days PD: Normal: number analyzed (Participants) | 30 | 28
  Temperature: 4th Inj,14 days PD: Normal | 30 | 28

ADVERSE EVENTS:
Time Frame: Baseline up to 24 weeks after last dose of treatment (Up to 300 weeks)
Description: Treatment emergent AEs are presented regardless of seriousness or relationship to investigational product.
Arm/Group | BIIB019
Serious Adverse Events (participants affected / at risk) | 148/410
Other Adverse Events (participants affected / at risk) | 296/410
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB019 (N=410)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 6
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Choroiditis (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 3
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Lip oedema (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Impaired healing (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Jaundice hepatocellular (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Hepatitis c (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Hiv infection (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Wound infection (Infections and infestations) | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Spinal column injury (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prolactinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 62
Neurological decompensation (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Glomerulonephritis (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephroptosis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Uterine inflammation (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Drug detoxification (Surgical and medical procedures) | 1
Eyelid operation (Surgical and medical procedures) | 1
Mammoplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB019 (N=410)
Lymphadenopathy (Blood and lymphatic system disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 25
Bronchitis (Infections and infestations) | 28
Nasopharyngitis (Infections and infestations) | 68
Pharyngitis (Infections and infestations) | 42
Respiratory tract infection viral (Infections and infestations) | 35
Upper respiratory tract infection (Infections and infestations) | 60
Urinary tract infection (Infections and infestations) | 42
Viral infection (Infections and infestations) | 23
Fall (Injury, poisoning and procedural complications) | 21
Alanine aminotransferase increased (Investigations) | 61
Aspartate aminotransferase increased (Investigations) | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 39
Headache (Nervous system disorders) | 44
Multiple sclerosis relapse (Nervous system disorders) | 110
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.